CLINICAL TRIAL: NCT00264017
Title: Palladium-103 Seed Implant and Single Daily Dosing of Uroxatral Vs Twice Daily Dosing of Flomax-A 3 Month Retrospective Efficacy Analysis
Brief Title: Palladium-103 Seed Implant and Single Daily Dosing of Uroxatral Vs. Twice Daily Dosing of Flomax- A 3 Month Retrospective Efficacy Analysis
Status: Completed | Type: Observational
Sponsor: Dattoli Cancer Center and Brachytherapy Research Institute (Other)
Collaborators: Sanofi (Industry)
Other Study IDs: L0087
Record Dates: First submitted 2005-12-06; First posted 2005-12-12 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 2005-11

CONDITIONS: Prostate Cancer Patients Undergoing External Radiation and Seed Implantation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
In the past ten years, newer drugs with more selective affinity for the alpha-receptor have been introduced. Alfuzosin (Uroxatral) and Tamulosin(Flomax are two second generation alpha-blockers. In the course of our clinical proctice, both drugs have been used routinely. This retrospective comparison is intended to be a priliminary comparison of their effectiveness and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Males age 45-80 years
* Diagnosis of prostate cancer
* Status post IMRT and Palladium-103 seed implantation and initiated alpha blocker therapy with alfuzosin10mg daily or tamulosin 0.4mg bid at time of seed implantation
* Baseline AUA score< or =12
* May be on antiandrogenand/or alpha reductase therapy
* Patients receiving IMRT followed by Palladium-103 Brachytherapy implantation as the primary therapy for prostate cancer with curatives intent -

Exclusion Criteria:

* History of insulin-dependent diabetes
* Uncontrolled hypertention
* History of symptomtic hypotension (including syncope and dizziness)
* Pre-existing obstructive uropathy based on history of BPH and or Acute Urinary Retention
* Pre-existing prostatitis either continuous or intermittent
* Concurrent use of any other anticholinergics
* previous or concurrent usage of LHRH agonist

Ages: 45 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Dattoli, MD, Principal Investigator — Dattoli Cancer Center and Brachytherapy Research Institute
Locations (1):
- Dattoli Cancer Center and Brachytherapy Research Institute, Sarasota, Florida, United States